CLINICAL TRIAL: NCT03848715
Title: Sleep and Healthy Aging Research on Depression for Younger Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Chloe Boyle, PhD, Postdoctoral Fellow, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16-000583-AM-00016
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Anhedonia; Depression
MeSH Terms: conditions — Anhedonia; Depression | interventions — Endotoxins

STUDY DESIGN:
Intervention Model Description: Endotoxin vs Placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinded infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endotoxin (Experimental): Endotoxin 0.8 ng/kg body weight; 1 infusion
  Interventions: Biological: Endotoxin
- Placebo (Placebo Comparator): same volume of 0.9% saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Endotoxin — Endotoxin
  Arms: Endotoxin
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Compelling evidence indicates inflammation plays a role in depression, but potential mechanisms linking inflammation to depression, such as dysregulated reward processing, are poorly understood. This study comprehensively evaluates effects of inflammation on reward across dimensions (e.g., anticipating versus receiving a reward) and types (e.g., money vs. smiling faces) in younger and older women. Characterizing how inflammation shapes the dynamic and multidimensional reward system, and how this may differ by age, may give insight into risk factors for depression and help identify critical points for intervention.

DETAILED DESCRIPTION:
This study will use an inflammatory challenge (i.e., endotoxin) to assess effects of inflammation on the behavioral response to social and non-social rewards, using tasks that assess reward motivation, sensitivity, and learning. Both elevated inflammation and reward dysregulation are associated with depression and have been shown to predict depression onset; understanding how inflammation alters the reward system in the laboratory setting may provide insight into risk factors and help identify potential areas for intervention. In this placebo-controlled, randomized, double-blind study of low dose endotoxin in 40 adult premenopausal women (25-44 y), the investigators will examine effects of endotoxin on reward responsiveness across dimensions (i.e., motivation, sensitivity, learning) and reward types (e.g., social and non-social). The investigators hypothesize that as compared to placebo, endotoxin will 1) decrease non-social reward responses across reward dimensions; 2) decrease "general" social reward responses across reward dimensions; 3) increase "close" social reward responses across reward dimensions; 4) decrease resting eye blink rate (EBR); EBR will be correlated with learning and motivation for non-social reward. The second component of the study is to examine whether effects of endotoxin on reward differ as a function of age; in particular it is hypothesized that effects will be more robust in younger compared to older women. In order to test for age differences, this study will use data from 40 older women (65+ y) participating in a parallel ongoing randomized controlled trial (ClinicalTrials.gov Identifier: NCT03256760). Thus, the investigation aims to: 1) Evaluate effects of inflammation on non-social reward as a function of age; 2) Evaluate effects of inflammation on general and close social reward as a function of age; 3) Examine changes in dopaminergic activity as a mechanism linking effects of inflammation on non-social reward processing as a function of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be required to be in good general health (as evaluated during the phone and in-person baseline session)
* Participants will be biologically female and premenopausal (as evaluated by self report).
* Participants will 25-44 years of age.

Exclusion Criteria:

* Presence of chronic mental or physical illness
* History of allergies, autoimmune, liver, or other severe chronic diseases,
* Current and regular use of prescription medications such as steroids, non-steroid anti-inflammatory drugs, aspirin, immune modifying drugs, opioid analgesics, statins, antihypertensive drugs, anti-arrhythmic drugs, and antidepressant medications (none in the last 6 months).
* Nightshift work or time zone shifts (> 3hrs) within the previous 6 weeks
* Previous history of fainting during blood draws.
* Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders;
* Presence of comorbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders;
* Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk;
* Presence of chronic infection, which may elevate proinflammatory cytokines;
* Presence of an acute infectious illness in the two weeks prior to an experimental session.
* Current Axis I psychiatric disorders as determined by the Research Version of the Structured Clinical Interview including a current major depressive disorder and substance dependence
* Lifetime history of suicide attempt or inpatient psychiatric admission.
* Current history of sleep apnea or nocturnal myoclonus; Phase-shift disorder, which will be identified by the Structured Clinical Interview and the Duke Structured Interview for Sleep Disorders
* Current smoking or excessive caffeine use (>600 mg/day) because of the known effects on proinflammatory cytokine levels;
* Evidence of recreational drug use from urine test.
* Body mass index > 35 because of the effects of obesity on proinflammatory cytokine activity
* Any clinically significant abnormality on screening laboratory tests
* Clinically significant abnormalities in electrocardiogram

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chloe C Boyle, PhD, Principal Investigator — University of California, Los Angeles; Michael R Irwin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Norman Cousins Center for Psychoneuroimmunology, University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyle CC, Cho JH, Eisenberger NI, Olmstead R, Sadeghi N, Castillo D, Irwin MR. Inflammation-induced depressed mood and reward responsivity as a function of age in female adults: a randomized controlled trial of endotoxin. Transl Psychiatry. 2025 Nov 26;16(1):6. doi: 10.1038/s41398-025-03752-2. PMID 41298372

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Clinical hold on LPS by FDA
Period: Overall Study
Arm/Group | Endotoxin | Placebo
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotoxin | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Full Range); unit: years] | 30 [25 to 41] | 35 [26 to 44] | 33 [25 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 14 | 18 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 8 | 11 | 19
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Non-social (Monetary) Reward Response (Reward Learning and Sensitivity)
Description: Implicit reward learning and sensitivity to monetary reward is assessed with the probabilistic reward task (PRT) a behavioral computer task; change in the magnitude of response bias from baseline to post-injection is the outcome measure. More positive response bias indicates a bias towards the more frequently reward stimuli (a better outcome); more negative response bias indicates a bias towards the less frequently reward stimuli (a worse outcome). This is not a standardized scale with minimum and maximum values. Response bias is calculated using a formula from signal detection theory and is a logarithmic ratio derived from choice frequencies. The formula is log b=1/2log((Rich-correct+.5) *(Lean-incorrect+.5)/(rich-incorrect+.5) * (lean-incorrect+.5)), where rich refers to the more frequently rewarded option and lean refers to the less frequently rewarded option.
Time Frame: Baseline and post-injection (2.25 hrs)
Population: For the Probabilistic Reward Task data are cleaned according to pre-specified quality controlled (QC) guidelines; data that do not meet these QC requirements are not included (e.g., participants who have accuracy less than 50%)
Measure: Mean (Standard Deviation); unit: response bias
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 14 | 17
response bias
  Baseline (pre-injection) PRT TASK | .563 (.292) | .307 (.409)
  Post-injection PRT TASK | .309 (.478) | .366 (.460)
Statistical Analysis 1: Comparison: Endotoxin vs Placebo; Test type: Superiority; p = .16, Regression, Linear

2. Primary Outcome: Non-social (Monetary) Reward Response (Reward Motivation)
Description: Motivation for monetary reward is assessed with a 10-minute version of the Effort Expenditure for Rewards Task (EEfRT), a behavioral computer task; change in the amount of hard trials chosen (relative to total trials) from baseline to post-injection is the outcome measure. The task is analyzed using generalized estimating equations (GEE) with a binary outcome; outcome values at each timepoint therefore range from 0 to 1, with higher numbers indicating higher motivation (a better outcome). The predictor for the GEE model is a time (coded as 0 and 1) by condition (coded as 0 and 1) interaction term. A negative result in the boxes below for each condition separately indicates a pre-to post-injection decrease in the proportion of hard trials chosen.
Time Frame: Baseline and post-injection (2.1 hrs)
Measure: Number (95% Confidence Interval); unit: Proportion of hard trials
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 18 | 22
Proportion of hard trials | -.3597425 [-.6121048 to -.1073803] | -.0876787 [-.2934619 to .1181044]

3. Primary Outcome: Non-social (Monetary) Reward Response (Reward Sensitivity)
Description: Sensitivity for monetary reward is assessed with a 10-minute version of the Effort Expenditure for Rewards Task (EEfRT) a behavioral computer task, tested as the strength of the association between increases in potential monetary reward for hard trials and selection of hard (vs) easy trials during the task. This is tested using generalized estimating equations, with condition (LPS vs. placebo) by time (pre vs post-injection) by reward magnitude (ranges from $1-$4.12) predicting hard (vs easy) trial choice. More positive values indicate higher reward sensitivity ( a better outcome), and lower values indicate lower reward sensitivity. The unit of measurement for the task is the proportion of hard trials chosen; the unit of measurement for the reward sensitivity outcome is a beta coefficient. For example, a positive coefficient for reward magnitude in the GEE output means that as the reward amount increases by one unit (e.g., $1), the odds of choosing the high-effort option increase.
Time Frame: Baseline and post-injection (2.1 hrs)
Measure: Number (95% Confidence Interval); unit: Proportion of hard trials chosen
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 18 | 22
Proportion of hard trials chosen | -.0525937 [-.1125722 to .0073848] | .0521303 [.0032571 to .1010036]

4. Primary Outcome: General Social Reward Response (Reward Sensitivity Via Emotional Dot Probe)
Description: Sensitivity to general social reward cues (i.e., response to positive emotional faces) assessed as positive attentional bias with an emotional dot probe task. Attentional bias is assessed by measuring reaction times to targets that appear in the same location as emotional (e.g., happy faces) versus neutral cues (e.g., neutral faces).
  Outcomes are change from baseline to post-injection in attentional bias towards positive vs neutral faces. Higher positive attentional bias scores indicate higher sensitivity to reward; negative attentional bias score indicate less sensitivity to reward. A score of 0 indicates no bias.
  The attentional bias score is derived by subtracting the reaction time in ms on congruent trials (dot replaces an emotional face) from the reaction time on incongruent trials (dot replaces the neutral face).
Time Frame: Baseline and post-injection (2.7 hrs)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 16 | 20
milliseconds | 11.85463 (18.61149) | 5.806407 (38.32138)

5. Primary Outcome: General Social Reward Response (Reward Sensitivity Via Face Morphing Task)
Description: Sensitivity to general social reward cues (i.e., response to positive emotional faces) assessed as positive emotion detection with a face morphing task. The outcome is the absolute change from baseline to post-injection in the percent of accurate responses. Higher accuracy is an indicator of higher sensitivity to reward and lower accuracy is an indicator of lower sensitivity to reward.
Time Frame: Baseline and post-injection (2.8 hrs)
Measure: Mean (Standard Error); unit: Percentage of accuracy
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 18 | 19
Percentage of accuracy | .0092593 (.0190538) | .0657895 (.0185456)

6. Primary Outcome: General Social Reward Response (Social Reward Motivation)
Description: Motivation for general social reward is assessed via self-report; participants rate their desire to engage in 3 different activities, one of which is social, on a 1 (not at all) to 10 (extremely) Likert scale.; change in desire for the social activity from baseline to post-injection is the outcome variable. Higher values indicate higher motivation.
Time Frame: Baseline and post-injection (2 hrs)
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 17 | 21
change in score on a scale | -2.94 (3.40) | -.29 (1.65)

7. Secondary Outcome: Depressed Mood Subscale of the Profile of Mood States (POMS)
Description: The Depressed Mood Subscale of the POMS is a self-reported assessment of depressed mood in which subjects rate severity of depressed mood using a visual analog scale from 1 to 10 (10 being most severe). Each timepoint is scored and analyses examine the temporal profile of change with assessment every hour. The outcome reported below is the mean score at 2-hours post-injection, which is when the response to endotoxin is known to peak. Higher values indicate more depressive symptoms.
Time Frame: Hourly, from pre-injection (T0) to 9 hours later (T9)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Endotoxin | Placebo
Number analyzed (Participants) | 18 | 22
score on a scale | 6.939871 (1.952918) | 2.680794 (1.762826)

8. Secondary Outcome: Close Social Reward Response
Description: Participants spend 5 minutes talking about a "close other" to a research assistant trained in reflective listening and provide ratings of current negative and positive emotion on visual analogue scales (0=not at all; 100=extremely) using items from the Profile of Mood States. Outcome variables are change in self-report positive emotion from pre to post-discussion, and percentage of positive and negative emotional words used during the discussion (scored with Linguistic Inquiry and Word Count Software). Higher positive emotion and higher percentage of positive words indicates a greater social reward response.
Time Frame: Post-injection (2.9 hrs)
Reporting Status: Not Posted, anticipated posting 2026-08

9. Secondary Outcome: Consummatory Daily Reward Response
Description: Participants indicate the extent to which they enjoyed 10 activities (social, non-social, close social) on a 0-100 visual analogue scale (0= not at all; 100=extremely) at five random times during the day; change in enjoyment in each of the domains from pre to post-experimental session is the outcome for consummatory reward. Higher values indicate higher reward response.
Time Frame: 14 days (7 days pre-injection; 7 days post-injection).
Reporting Status: Not Posted, anticipated posting 2026-07

10. Secondary Outcome: Dopaminergic Activity
Description: Count of eye blinks (resting eye blink rate; EBR) over a five minute period; the outcome is change in EBR from pre to post-injection. Higher values indicate higher dopaminergic activity.
Time Frame: Baseline and post-injection (1.9 hrs)
Reporting Status: Not Posted, anticipated posting 2026-07

11. Secondary Outcome: Anticipatory Daily Reward Response
Description: Participants rate how much they are currently looking forward to different categories of rewarding activities on an analogue scale (0= not at all; 100=extremely); change from pre to post-experimental session is the outcome for anticipatory reward. Higher values indicate higher reward response.
Time Frame: 14 days (7 days pre-injection; 7 days post-injection).
Reporting Status: Not Posted, anticipated posting 2026-07

12. Other Pre Specified Outcome: Negative Emotion Regulation Capacity
Description: Participants complete a 30 minute standardized emotion regulation task that includes two phases: a reactivity phase and a regulation phase, and assesses the ability to down-regulate negative emotional response to standardized images, using instructed reappraisal strategies. The dependent variable is the degree to which self-reported emotion changes when reacting to versus reappraising emotion stimuli. Participants rate how negative they feel on a 0 (not at all) to 100 (extremely) visual analogue scale before and after film clips. The change in negative emotion when reacting is compared to the change in negative emotion when regulating. More positive values indicate better emotion regulation.
Time Frame: post-injection (approximately 3 hrs)
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 10 hour period for each participant.
Arm/Group | Endotoxin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03848715/Prot_SAP_001.pdf